CLINICAL TRIAL: NCT03735368
Title: Dexmedetomidine With or Without Pregabalin Premedication for Conscious Sedation During Cataract Surgery Under Topical Anesthesia. A Randomized Double-blind Placebo-controlled Trial.
Brief Title: Dexmedetomidine and Pregabalin for Conscious Sedation During Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abd-Elazeem Abd-Elhameed Elbakry (Other)
Responsible Party: Sponsor-Investigator, Abd-Elazeem Abd-Elhameed Elbakry, assistant professor, Menoufia University
Organization: Menoufia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/10/15/5
Record Dates: First submitted 2018-11-04; First posted 2018-11-08 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Dexmedetomidine; Pregabalin; Anesthesia; benoxinate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, the surgeons and the research team will be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): placebo oral capsule+ dexmedetomidine+topical anesthesia
  Interventions: Drug: Dexmedetomidine Injection; Drug: Placebo oral capsule; Drug: topical anesthesia
- Dexmedetomidine- Pregabalin (Active Comparator): Pregabalin Oral Capsule +Dexmedetomidine Injection+topical anesthesia
  Interventions: Drug: Dexmedetomidine Injection; Drug: Pregabalin Oral Capsule; Drug: topical anesthesia

INTERVENTIONS:
Drug: Dexmedetomidine Injection — Dexmedetomidine Injection 1 μg/kg then 0.5-1 μg/kg/h infusion
  Other Names: Dexmedetomidine
Drug: Placebo oral capsule — placebo oral capsules
  Other Names: placebo
  Arms: Control
Drug: Pregabalin Oral Capsule — 150 mg pregabalin Oral Capsule
  Other Names: pregabalin
  Arms: Dexmedetomidine- Pregabalin
Drug: topical anesthesia — topical anesthesia of the eye by Benoxinate Hydrochloride 0.4% Eye Drops
  Other Names: Benoxinate Hydrochloride 0.4% Eye Drops

SUMMARY:
Although topical anesthesia by eye drops for cataract surgery is a non-invasive technique but it may provide insufficient anesthesia which requires the intraoperative use of additional topical local anesthetics and raises the need for sedation.

DETAILED DESCRIPTION:
The present study is constructed to evaluate the effect of pregabalin on sedation using dexmedetomidine for cataract surgery under topical anesthesia . In the dexmedetomidine-pregabalin group, the patients will be premedicated by pregabalin. In the placebo group (control group) the patients will be premedicated by placebo capsules. All patients will be sedated by dexmedetomidine. Sedation will be assessed as a primary outcome measurement where pain, vital signs, intraoperative and postoperative pain, total analgesic needs and side effects will be assessed as secondary outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* American Society Of Anesthesiologists (ASA) I and II physical status.
* Scheduled for cataract extraction under topical anesthesia.

Exclusion Criteria:

* Hepatic or renal impairment.
* Taking chronic psychotropic medications.
* Mental instability.
* Morbid obesity.
* Alcohol abuse.
* Substance abuse.
* Pregnant and lactating females.
* History of allergy to the study drugs used

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
sedation score changes | baseline,1hour after premedication, intraoperative every 5 minutes ,postoperative every 6hours for 24 hours
  Ramsay sedation score from 1 to 6. score 2 to 4 is acceptable sedation. Score 5 or 6 is excessive sedation.

SECONDARY OUTCOMES:
pain score changes | baseline,1hour after premedication, intraoperative every 5 minutes ,postoperative every 6hours for 24 hours
  verbal pain score (VPS) from 0 = no pain to 10= the worst pain imaginable. scor ≥ 3 indicates need of analgesia
heart rate changes | baseline,1hour after premedication, intraoperative every 5 minutes ,postoperative every 6hours for 24 hours
  beats/minute
arterial blood pressure changes | baseline,1hour after premedication, intraoperative every 5 minutes ,postoperative every 6hours for 24 hours
  mmHg
arterial oxygen saturation | baseline,1hour after premedication, intraoperative every 5 minutes ,postoperative every 6hours for 24 hours
  the percentage of hemoglobin saturation with oxygen in arterial blood.
respiratory rate | baseline,1hour after premedication, intraoperative every 5 minutes ,postoperative every 6hours for 24 hours
  breath/minute
total dexmedetomidine consumption | intraoperatively
  ug
Incidence of respiratory depression | from administering premedication till 24 hours postoperative.
  percentage
Incidence of hypotension | from administering premedication till 24hours postoperative
  percentage
Incidence of bradycardia | from administering premedication till 24hours postoperative
  percentage
Incidence of ataxia | from administering premedication till 24hours postoperative
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, MD, Principal Investigator — Assistant professor
Locations (1):
- Faculty of Medicine, Cairo, Shebin El-kom, Egypt